CLINICAL TRIAL: NCT06656299
Title: Evaluation of Post-Operative Analgesic Efficacy of Bilateral External Oblique Intercostal Plane Block Versus Wound Site Infiltration Control Group in Patients Underwent Laparoscopic Cholecystectomy Surgery
Brief Title: EOIB for Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOIB
Record Dates: First submitted 2024-10-20; First posted 2024-10-24 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Cholecystitis; Cholecystitis, Acute; Cholecystitis, Chronic; Cholecystitis; Gallstone
Keywords: External Oblique Intercostal Plan Block; Wound Infiltration; Laparoscopic Cholecystectomy; Postoperative pain
MeSH Terms: conditions — Cholecystitis; Cholecystitis, Acute; Bronchiolitis Obliterans Syndrome; Gallstones; Pain, Postoperative | interventions — Bupivacaine; Anesthetics, Local; Acetaminophen; Tramadol; Ondansetron

STUDY DESIGN:
Intervention Model Description: There are two groups for this study
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and outcomes assessor wil be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup E (External Oblique Intercostal Plane Block) (Active Comparator): At the end of the surgical procedure,a high-frequency linear probe will be sterilely covered,and an 80mm block needle will be used for the procedure.Under sterile conditions,the ultrasound probe will be placed in a parasagittal position in the area between the anterior axillary line and the midclavicular line at the level of the 10th rib, and then slid cranially along the longitudinal axis to the level of the 6th and 7th ribs. After visualizing the external oblique muscle, the block needle will be inserted using an in-plane technique,and 5ml of saline will be administered to confirm the location at the external oblique intercostal plane between the external oblique muscle and the 6th rib. Once the location is confirmed, 20cc of 0.25%bupivacaine will be infiltrated into the EOIP. The same procedure will be applied to the opposite side (totally 40 ml).
  Interventions: Device: ultrasound guided external oblique intercostal plane block; Drug: paracetamol, tramadol, and ondansetron
- Grup T ( Trocar entry site infiltration) (Other): After the trocar removed during the surgical procedure, the surgeon will administer 5 ml of 0.25% bupivacaine infiltration to each trocar entry site.
  Interventions: Drug: Bupivacaine injection; Drug: paracetamol, tramadol, and ondansetron

INTERVENTIONS:
Device: ultrasound guided external oblique intercostal plane block — ultrasound guided external oblique intercostal plane block
  Arms: Grup E (External Oblique Intercostal Plane Block)
Drug: Bupivacaine injection — 5 ml local anesthetic for each trocar sides
  Other Names: Local anesthetic injection
  Arms: Grup T ( Trocar entry site infiltration)
Drug: paracetamol, tramadol, and ondansetron — As standard multimodal analgesia, 20 min before the end of the surgery patients will receive 1 g of paracetamol, 1-2 mg/kg of tramadol, and 4 mg of ondansetron via intravenous infusion.
  All patients will be recovered in the PACU, and after confirming an Aldrete score of >9, a PCA (patient-controlled analgesia) device will be installed with morphine prepared at a dose appropriate for the patient's age. Patients will be administered paracetamol 1 gr IV every 8 hours in the postoperative period. When patients have a Numerical Rating Scale (NRS) score is ≥ 4, 1 mg/kg iv tramadol will be administered as a rescue analgesic

SUMMARY:
Laparoscopic cholecystectomy, while less painful compared to conventional methods, is still a surgery that can cause significant pain for patients. Preventing postoperative pain is crucial for reducing respiratory complications, shortening hospital stays, and increasing patient satisfaction. Interfascial plane blocks have been widely used for postoperative analgesia in recent years worldwide. The External Oblique Intercostal Plane Block is one of the interfascial plane blocks used in abdominal surgeries. In our study, we aimed to compare the postoperative pain scores of patients who underwent laparoscopic cholecystectomy under general anesthesia, specifically between those who received the external oblique intercostal plane block and those who had trocar entry site infiltration.

DETAILED DESCRIPTION:
Despite the advancements in surgical and anesthesia techniques, pain following surgical interventions remains a significant issue concerning patient health and comfort today. The physiological response resulting from surgical trauma and stress can lead to various unwanted conditions in the pulmonary, cardiovascular, gastrointestinal, metabolic, and neuroendocrine systems. These complications negatively impact wound healing, length of hospital stay, and costs. The primary goal in managing pain after surgery is to facilitate the healing process, avoid potential side effects associated with analgesic treatments, and enhance patient comfort.

Cholecystectomy, which plays a significant role among abdominal surgical interventions, can currently be performed using two distinct techniques: open and laparoscopic.

Laparoscopic cholecystectomy is considered the gold standard treatment for symptomatic cholelithiasis due to its ability to cause less trauma compared to open surgery, facilitate faster recovery in patients, result in less postoperative pain, and allow patients to return to their normal lives more quickly.

There are three components of postoperative pain observed after laparoscopic cholecystectomy. These include somatic pain associated with the laparoscopic trocar entry incisions in the anterior abdominal wall, visceral pain due to pneumoperitoneum and surgical dissection of the gallbladder, and referred shoulder pain resulting from the stimulation of the phrenic nerve by residual carbon dioxide gas.

Effective management of postoperative pain is crucial for reducing respiratory complications, shortening hospital stay, and increasing patient satisfaction. In this context, both nonsteroidal intravenous analgesics and opioids are used. However, opioids have undesirable side effects, including respiratory depression, nausea and vomiting, and reduced gastrointestinal motility. Therefore, multimodal analgesia methods that combine intravenous analgesics with regional anesthesia are preferred, allowing for the reduction of drug-related side effects while providing safe and effective postoperative analgesia.

Interfascial plane blocks have been widely used for postoperative analgesia worldwide in recent years. When using long-acting local anesthetics and performed under ultrasound guidance, peripheral nerve blocks can be administered more easily, effectively, and reliably, providing analgesia for approximately 8 to 24 hours.

The External Oblique Intercostal Plane Block (EOIB) is one of the interfascial blocks used in upper abdominal surgeries. The local anesthetic is administered between the anterior axillary line and the midclavicular line, specifically in the fascia between the external oblique muscle and the sixth rib. Cadaver studies have demonstrated the spread of local anesthesia to the anterior cutaneous nerve at the T6-9 dermatomes and to the lateral cutaneous nerve at the T6-10 dermatomes. These studies suggest that the EOIB could be part of multimodal analgesia in upper and lateral abdominal surgeries. In this study, our hypothesis is that the EOIB may reduce the amount of opioids used in postoperative pain management, decrease opioid-related side effects, enhance patient comfort, and shorten the recovery process.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 who will be scheduled for an elective laparoscopic cholecystectomy under general anesthesia
* ASA (American Society of Anesthesiologists) I-II-III

Exclusion Criteria:

* presence of coagulation disorder
* infection at the injection site of the block
* known allergy to local anesthetics
* advanced hepatic, heart or renal failure
* history of abdominal surgery or trauma
* conversion of laparoscopic to open surgery
* consumption of any pain killers within the 24 h before the operation
* chronic opioid consumption
* pregnancy
* alcohol or drug abuse
* body mass index (BMI) ≥ 35 kg m-2
* Impairment of the patient's cognitive functions (such as Alzheimer's disease, dementia, etc.).
* Cholecystectomy cases performed under emergency conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
NRS (Numeric Rating Skore) | Postoperative 24 hours
  The primary outcome variable is Numerical Rating Scale scores both at rest and motion. A blinded anesthesiologist will assess postoperative pain during rest and motion at the postoperative 15th,30th and 60th minute, second,6th, 12th and 24th hour by using 11-point Numerical Rating Scale which ranges from '0' (means no pain) to '10' (means worst pain imaginable).

SECONDARY OUTCOMES:
Opioid Consumption | Postoperative 24 hours
  First 24 hours total morphine consumption with patient controlled analgesia
Time to first rescue analgesic | Postoperative 24 hours
  The time for administration of first rescue analgesic.
Adverse Events | Postoperative 24 hours
  Incidence of nausea and vomiting during postoperative 24 hour time period will be noted.
Metoclopromide Consumption | Postoperative 24 hours
  The severity of the nausea will be assessed on a 4 -point scale (0=none 1=mild, 2=moderate 3=severe). If the patients nausea score is ≥2 the patient will receive 10 mg metoclopromide.
Quality of recovery levels between groups by using QoR-15 questionnaire | Postoperative 24 hours
  A 15-parameter Quality of Recovery score (QoR-15) has been recommended as the optimum tool to evaluate overall patient-centers measures of recovery after surgery, including pain. It is a questionnaire that is given to patients to do postoperatively and is scored from 0 to 150 where 150 indicates that the patient has had an excellent recovery QoR-15 score will be recorded on the morning of operation and at the postoperative 24th hour

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not share IPD

REFERENCES:
- [Background] Korkusuz M, Basaran B, Et T, Bilge A, Yarimoglu R, Yildirim H. Bilateral external oblique intercostal plane block (EOIPB) in patients undergoing laparoscopic cholecystectomy: A randomized controlled trial. Saudi Med J. 2023 Oct;44(10):1037-1046. doi: 10.15537/smj.2023.44.10.20230350. PMID 37777270
- [Background] Doymus O, Ahiskalioglu A, Kaciroglu A, Bedir Z, Tayar S, Yeni M, Karadeniz E. External Oblique Intercostal Plane Block Versus Port-Site Infiltration for Laparoscopic Sleeve Gastrectomy: A Randomized Controlled Study. Obes Surg. 2024 May;34(5):1826-1833. doi: 10.1007/s11695-024-07219-z. Epub 2024 Apr 2. PMID 38565828
- [Background] Mehmet Selim C, Halide S, Erkan Cem C, Onur K, Sedat H, Senem U. Efficacy of Unilateral External Oblique Intercostal Fascial Plane Block Versus Subcostal TAP Block in Laparoscopic Cholecystectomy: Randomized, Prospective Study. Surg Innov. 2024 Aug;31(4):381-388. doi: 10.1177/15533506241256529. Epub 2024 May 23. PMID 38780355